CLINICAL TRIAL: NCT02781376
Title: Evidence-based Diagnosis and Management of Pediatric Obstructive Sleep Apnea in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other); American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Sarah Honaker, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1603153280; 2015 (Other Grant/Funding Number: American Sleep Medicine Foundation)
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Primary Care; Computer Decision Support System; Guidelines; Snoring
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHICA-OSA (Experimental): Two clinics will be randomized to receive the advanced CHICA-OSA computer decision support system designed to support PCPs in evidence-based identification and management of pediatric OSA. This module includes a snoring identification component (received by the control group).
  Interventions: Other: CHICA OSA
- Control (Other): Two clinics will be randomized to receive a control computer decision support system module that automates screening for snoring and alerts the PCP, but does not provide any additional guidance on evidence-based diagnosis or management.
  Interventions: Other: Snoring Identification Only

INTERVENTIONS:
Other: CHICA OSA — Computer decision support system module that assesses snoring, assesses additional OSA symptoms, provides guideline-based recommendation to PCPs, and reassesses for residual OSA symptoms.
  Arms: CHICA-OSA
Other: Snoring Identification Only — Computer decision support system module that assesses snoring and alerts the PCP when caregivers endorse snoring.
  Arms: Control

SUMMARY:
Obstructive Sleep Apnea (OSA) is prevalent in children and adolescents and associated with a variety of negative consequences affecting health and cognitive functioning. While clinical guidelines outline effective strategies for the diagnosis and management of pediatric OSA, rates of screening, identification, and management in primary care settings remain low. The aim of the current study is to evaluate the use of a computer decision support system module (CHICA-OSA) designed to improve adherence to OSA guidelines in pediatric primary care clinics. All children ages 1-11 years will be screened for snoring and other symptoms of OSA in the waiting room prior to a visit to their primary care provider (PCP). In clinics randomly assigned to CHICA-OSA, caregivers of snoring children will report on additional OSA symptoms, and PCPs will receive automated prompts in the electronic health record (EHR) to provide evidence-based evaluation and appropriate referral for testing. For children sent for polysomnography (PSG), PCPs will receive automated prompts to reassess symptoms at the next visit. We hypothesize that clinics using CHICA-OSA will have better adherence to guidelines, as evidenced by higher rates of identifying OSAS, referral for PSG, and re-assessment following treatment.

DETAILED DESCRIPTION:
Study Design: This study will use a cluster randomized control trial (RCT) over a two-year period in four pediatric community clinics affiliated with our institution. To minimize contamination, randomization will occur by clinic, with the individual patient as the unit of analysis. Four clinics are already matched in pairs to facilitate a balance of patient numbers and demographics, and a coin flip will determine which clinic pair will receive CHICA-OSA and which will serve as control clinics. The two control clinics also have the CHICA system in place but the only intervention pertaining to sleep will be a simple module that identifies snoring children. While receiving automated prompts to help identify snoring children, PCPs in control clinics will evaluate and manage OSA using their standard methods (i.e., treatment-as-usual).

Participants: Participants will include all children between the ages of 1 and 11 years presenting to their PCP to one of four pediatric community clinics located in Indianapolis, Indiana.

CHICA System: CHICA is comprised of: (1) a knowledge base of pediatric guideline rules; (2) a repository of patient data; (3) a tablet user interface; and (4) an interface to the existing electronic medical record system. The result is a system that both delivers "just-in-time" patient-relevant guidelines to PCPs during the clinical encounter and captures accurate structured data from all who interact with it. In the waiting room caregivers complete a prescreening form (PSF), available in English and Spanish, consisting of a series of twenty surveillance questions tailored to the child's age and past history. A positive response to a question may trigger additional follow-up questions. During the clinic visit, relevant feedback from caregiver responses and information about clinical guidelines are displayed prominently on a provider worksheet (PWS) in the electronic health record.

Visit 1. While in the waiting room, caregivers for all eligible children will respond to an item on the PSF as follows: "Does your child consistently snore 3 or more nights per week?" For caregivers in CHICA-OSA clinics, a "yes" response will trigger additional questions about signs and symptoms of OSA. Specific items corresponding to the symptoms will be taken from the Pediatric Sleep Questionnaire (PSQ19) and include observed apnea, snorts, gasps, daytime sleepiness, and other signs and symptoms listed in the AAP guideline paper. The PCP will then receive a PWS prompt listing signs and symptoms that apply to the child, based on either existing data in the electronic record (e.g., current ADHD diagnosis; overweight) or on caregiver responses to items assessed in the waiting room (e.g., observed apnea; daytime sleepiness). When evidence-based criteria are met, according to the 2012 American Academy of Pediatrics (AAP) guidelines, the PCP will be encouraged to refer the child (for a PSG, to a sleep specialist, or to an ENT).

In the control clinics, parents will complete a surveillance question about snoring, and PCPs will receive a generic prompt but will not receive any additional information about signs and symptoms or guidance on how to further evaluate or manage. For children in both the CHICA-OSA and control clinics, if a caregiver does not report snoring the item about snoring will be repeated one year later.

Subsequent Visits: At the next visit (sick or WCC), snoring will again be assessed as one of the health surveillance questions for all eligible children. However, children from the CHICA-OSA clinics who were referred for PSG at the previous visit will receive an additional item asking whether or not the child has had an adenotonsillectomy in the past year. If the child has not had this surgery the PCP will receive a prompt to assess the outcome of the original referral (e.g., PSG did not suggest OSA; PSG suggested OSA and surgery scheduled; PSG scheduled; adenotonsillectomy scheduled; family does not have appointment) and re-refer if appropriate. If a caregiver reports that a child has had a T&A and no longer snores, the PCP will not receive any additional prompts and snoring will be reassessed in two years. However, if a caregiver reports residual snoring after surgery, the provider will receive a prompt to refer for possible residual OSA.

Collaborators on this study include: Stephen Downs, MD, Indiana University School of Medicine; Ameet Daftary, MD, Indiana University School of Medicine; and Tamara Dugan, MS, Indiana University School of Medicine

ELIGIBILITY:
Inclusion Criteria:

* Children between 1-11 years seen at one of four participating primary care clinics in Indianapolis, Indiana.
* Caregiver completes screening items.

Exclusion Criteria:

* None

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Rate of Appropriate Referral | Within 6 months of the date at which snoring was first identified
  Appropriate referral is defined as children with snoring and at least one additional OSA sign or symptom who were referred by the PCP to PSG, ENT, or Sleep Specialist. The number of appropriate referrals will be divided by the number of children identified by the CHICA system as snoring. This outcome will be compared between control and intervention clinics.

SECONDARY OUTCOMES:
Rate of Confirmed OSA | Day of the PSG (assessed through study completion, up to 18 months)
  Number of children receiving an confirmed OSA diagnosis (apnea hypopnea index 1.5 or greater) by PSG. This number will be divided by the number of children referred to PSG through CHICA who completed a PSG. Rate will be compared between the intervention and control clinics.
Rate of Completed PSG | Within 6 months of the date child was refered for PSG
  Number of completed PSGs amongst those referred for PSG through the CHICA system. Rate will be compared between intervention and control clinics.
Rate of Assessment for Residual OSA | Within 3 months of the first visit to the PCP after initiation of OSA treatment
  Rate of provider documentation of screening for snoring amongst those receiving OSA treatment (e.g., adenotonsillectomy, nasal steroid spray).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Honaker, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Honaker SM, Street A, Daftary AS, Downs SM. The Use of Computer Decision Support for Pediatric Obstructive Sleep Apnea Detection in Primary Care. J Clin Sleep Med. 2019 Mar 15;15(3):453-462. doi: 10.5664/jcsm.7674. PMID 30853049